CLINICAL TRIAL: NCT01188577
Title: Epinephrine Inhalation Aerosol USP, an HFA-MDI CLINICAL STUDY-B2 FOR ASSESSMENT OF PHARMACOKINETICS (A Randomized, Evaluator-Blind, Single-Dose, Two Arm, Crossover, PK Study in Healthy Volunteers)
Brief Title: Epinephrine Inhalation Aerosol USP, a HFA-MDI Study for Assessment of Pharmacokinetics
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Amphastar Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: API-E004-CL-B2
Record Dates: First submitted 2010-08-24; First posted 2010-08-25 (Estimated); Results first posted 2014-10-24 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-06

CONDITIONS: Asthma; Bronchospasm; Wheezing; Shortness of Breath
Keywords: asthma; bronchospasm; wheezing; shortness of breath
MeSH Terms: conditions — Asthma; Bronchial Spasm; Respiratory Sounds; Dyspnea | interventions — Inhalation; Epinephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Epinephrine Inhalation Aerosol, HFA (Experimental): Experimental treatment of 10 inhalations of 125 mcg epinephrine base propelled by HFA 134a
  Interventions: Drug: Epinephrine Inhalation Aerosol, HFA
- Epinephrine Inhalation Aerosol, CFC (Active Comparator): Epinephrine Inhalation Aerosol, CFC propelled, 220 mcg/inhalation , 10 inhalations
  Interventions: Drug: Epinephrine Inhalation Aerosol

INTERVENTIONS:
Drug: Epinephrine Inhalation Aerosol, HFA — 10 inhalations of epinephrine inhalation aerosol, 125 mcg/inhalation
  Other Names: HFA epinephrine inhalation aerosol, 125 mcg/inhalation
  Arms: Epinephrine Inhalation Aerosol, HFA
Drug: Epinephrine Inhalation Aerosol — Epinephrine Inhalation Aerosol, 220 mcg/ inhalation, 10 inhalations
  Other Names: Primatene Mist; Epinephrine Inhalation Aerosol, USP
  Arms: Epinephrine Inhalation Aerosol, CFC

SUMMARY:
This study examines the pharmacokinetic profile of Armstrong's proposed Epinephrine Inhalation Aerosol USP, an HFA-MDI (E004), using a stable isotope deuterium-labeled epinephrine (epinephrine-d3) to differentiate the administered drug from the endogenous epinephrine, in healthy male and female adult volunteers. The current study is designed for a more thorough evaluation of the E004 Pharmacokinetics. Safety of E004 will also be evaluated, under augmented dose conditions.

DETAILED DESCRIPTION:
E004 is formulated with epinephrine free base as the active ingredient, and hydrofluoroalkane (HFA-134a) as the propellant.

In order to differentiate the inhaled epinephrine from the fluctuating background of endogenous epinephrine 1, a stable-isotope deuterium (2H) labeled epinephrine (epinephrine-d3) preparation will be used to formulate E004 inhalers, denoted as E004-d3. PK of E004 at 125 mcg of epinephrine-d3 per inhalation, will be compared to that of the currently marketed, non-labeled, Epinephrine-CFC MDI as the Reference Control (220 mcg per inhalation).

This study is a randomized, evaluator-blind, single dose, two-arm, crossover, PK study, to be conducted in ~18 healthy, male and female, adult volunteers. PK will be studied using E004-d3 at 125 mcg per inhalation (Arm T). A currently marketed, non-labeled, Epinephrine CFC-MDI will be used as a Reference Control (Arm C).

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy at screening;
* No clinically significant respiratory, cardiovascular and other systemic or organic illnesses;
* Body weight ≥ 50 kg for men and ≥ 45 kg for women,
* Sitting blood pressure ≤ 135/90 mm Hg;
* Demonstrating negative HIV, HBsAg and HCV-Ab screen tests;
* Women of child-bearing potential must be non-pregnant, non-lactating, and practicing a clinically acceptable form of birth control;
* Properly consented
* Other criteria apply

Exclusion Criteria:

* A smoking history of ≥10 pack-years, or having smoked within 6 months;
* Upper respiratory tract infections within 2 wk, or lower respiratory tract infection within 4 wk, prior to Screening;
* Any current or recent respiratory conditions that might significantly affect pharmacodynamic response to the study drugs;
* Known intolerance or hypersensitivity to the study MDI ingredients;
* Having been on other investigational studies, or donated blood, in the last 30 days;
* Other Criteria Apply

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2010-08; Primary Completion 2010-09 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Amphastar Pharmaceuticals, Inc.
Locations (1):
- Amphastar Site 0035, Cypress, California, United States

REFERENCES:
- [Background] Pinnas JL, Schachtel BP, Chen TM, Roseberry HR, Thoden WR. Inhaled epinephrine and oral theophylline-ephedrine in the treatment of asthma. J Clin Pharmacol. 1991 Mar;31(3):243-7. doi: 10.1002/j.1552-4604.1991.tb04969.x. PMID 2019665
- [Background] Hendeles L, Marshik PL, Ahrens R, Kifle Y, Shuster J. Response to nonprescription epinephrine inhaler during nocturnal asthma. Ann Allergy Asthma Immunol. 2005 Dec;95(6):530-4. doi: 10.1016/S1081-1206(10)61014-9. PMID 16400891
- [Background] Warren JB, Doble N, Dalton N, Ewan PW. Systemic absorption of inhaled epinephrine. Clin Pharmacol Ther. 1986 Dec;40(6):673-8. doi: 10.1038/clpt.1986.243. PMID 3780129
- [Background] Cripps A, Riebe M, Schulze M, Woodhouse R. Pharmaceutical transition to non-CFC pressurized metered dose inhalers. Respir Med. 2000 Jun;94 Suppl B:S3-9. PMID 10919679
- [Background] Dickinson BD, Altman RD, Deitchman SD, Champion HC. Safety of over-the-counter inhalers for asthma: report of the council on scientific affairs. Chest. 2000 Aug;118(2):522-6. doi: 10.1378/chest.118.2.522. PMID 10936150
- [Background] Simons FE, Gu X, Johnston LM, Simons KJ. Can epinephrine inhalations be substituted for epinephrine injection in children at risk for systemic anaphylaxis? Pediatrics. 2000 Nov;106(5):1040-4. doi: 10.1542/peds.106.5.1040. PMID 11061773
- [Background] Kushner DJ, Baker A, Dunstall TG. Pharmacological uses and perspectives of heavy water and deuterated compounds. Can J Physiol Pharmacol. 1999 Feb;77(2):79-88. PMID 10535697
- [Background] Bondesson E, Friberg K, Soliman S, Lofdahl CG. Safety and efficacy of a high cumulative dose of salbutamol inhaled via Turbuhaler or via a pressurized metered-dose inhaler in patients with asthma. Respir Med. 1998 Feb;92(2):325-30. doi: 10.1016/s0954-6111(98)90116-0. PMID 9616533
- [Derived] Kerwin EM, Marrs T, Luo MZ, Zhang JY. Pharmacokinetic Study of Epinephrine Hydrofluoroalkane (Primatene MIST) Metered-Dose Inhaler. J Aerosol Med Pulm Drug Deliv. 2020 Oct;33(5):282-287. doi: 10.1089/jamp.2019.1577. Epub 2020 May 18. PMID 32423275

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from a specialty clinic in Cypress, CA between 08/19/2010 and 09/09/2010.
Pre-assignment Details: A total of 35 subjects were screened, 23 subjects passed screening, consented and were randomized for participation in the study.
Groups:
- C, T: Subjects received one of the two treatments during each study visit, separated by a washout period of 3-14 days. Visit 1: Treatment C: Ten (10) inhalations of Epinephrine CFC-MDI (220 mcg/inhalation), totaling 2.20 mg of epinephrine, in 5 min; Visit 2: Treatment T: Ten (10) inhalations of E004 (125 mcg/inhalation), totaling 1.25 mg of epinephrine, in 5 min.
- T, C: Subjects received one of the two treatments during each study visit, separated by a washout period of 3-14 days. Visit 1: Treatment T: Ten (10) inhalations of E004 (125 mcg/inhalation), totaling 1.25 mg of epinephrine, in 5 min; Visit 2: Treatment C: Ten (10) inhalations of Epinephrine CFC-MDI (220 mcg/inhalation), totaling 2.20 mg of epinephrine, in 5 min.
Period: Visit 1
Arm/Group | C, T | T, C
Started | 11 | 12
Completed | 11 | 12
Not Completed | 0 | 0
Period: 3-14 Day Washout
Arm/Group | C, T | T, C
Started | 11 | 12
Completed | 11 | 12
Not Completed | 0 | 0
Period: Visit 2
Arm/Group | C, T | T, C
Started | 11 | 12
Completed | 11 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | C, T | T, C | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Continuous [Mean (Standard Deviation); unit: Years] | 22.8 (2.99) | 24.8 (2.93) | 23.8 (3.05)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 10 | 12 | 22
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 9 | 8 | 17
Region of Enrollment [Number; unit: participants]
  United States | 11 | 12 | 23

OUTCOME MEASURES:

1. Primary Outcome: Baseline Concentration (C0) of Total Epinephrine
Description: Patient PK blood samples were taken from a vein in a hand or arm via indwelling heparin-anticoagulated IV catheters, or by venipunctures at Baseline (prior to dosing) in each treatment period following a specified washout period (3-14 days), and were analyzed using an established analysis method. Baseline concentration (C0) is the concentration of epinephrine measured in the plasma at this time point.
Time Frame: 0 to 30 minutes prior to dosing
Population: Patients who: 1) have taken the valid pre-dose baseline PK sample 2) have correctly taken the randomized study drug treatment 3) have at least three of the four post-dose PK measurement btwn 2 and 10 min post-dose available and 4) have a minimum of twelve of the fifteen post-dose PK measurements for the entire 6 hour post-dose PK sampling period.
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Treatment T: Ten (10) inhalations of E004 (125 mcg/inhalation), totaling 1.25 mg of epinephrine, in 5 min
- Treatment C: Ten(10) inhalations of Epinephrine CFC-MDI (220 mcg/inhalation), totaling 2.20 mg of epinephrine, in 5 min
Arm/Group | Treatment T | Treatment C
Number analyzed (Participants) | 23 | 23
pg/mL | 2.6 (8.7) | 4.3 (16.7)

2. Primary Outcome: Peak Concentration (Cmax) of Total Epinephrine From Time Zero to 6 Hours Post-dose
Description: Patient PK blood samples were taken from a vein in a hand or arm via indwelling heparin-anticoagulated IV catheters, or by venipunctures at 0 (baseline), 2, 5, 7.5, 10, 12.5, 15, 20, 25, 30, 45, 60, 90, 120, 240, and 360 minutes post-dose in each treatment period and were analyzed using an established analysis method. Peak (maximum) concentration (Cmax) is the highest concentration of epinephrine measured in plasma during the treatment period.
Time Frame: Pre-dose to 6 hours post-dose
Population: Patients who: 1) have taken the valid pre-dose baseline PK sample 2) have correctly taken the randomized study drug treatment 3) have at least three of the four post-dose PK measurements btw 2 and 10 min post-dose available and 4) have a minimum of twelve of the fifteen post-dose PK measurements for the entire 6 hour post-dose PK sampling period.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Treatment T | Treatment C
Number analyzed (Participants) | 23 | 23
pg/mL | 862 (527) | 190 (119)

3. Primary Outcome: Area Under the Curve From Time Zero to 6 Hours Post-dose (AUC[0-6]) for Total Epinephrine
Description: Patient PK blood samples were taken from a vein in a hand or arm via indwelling heparin-anticoagulated IV catheters, or by venipunctures at 0 (baseline), 2, 5, 7.5, 10, 12.5, 15, 20, 25, 30, 45, 60, 90, 120, 240, and 360 minutes post-dose in each treatment period and were analyzed using an established analysis method. Area under the curve from time zero to 6 hours post-dose (AUC[0-6]) was calculated using the trapezoidal rule.
Time Frame: Pre-dose to 6 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pg*min/mL
Arm/Group | Treatment T | Treatment C
Number analyzed (Participants) | 23 | 23
pg*min/mL | 8498 (5213) | 6191 (4108)

4. Primary Outcome: Time to Reach Peak Concentration (Tmax) for Total Epinephrine
Description: Patient PK blood samples were taken from a vein in a hand or arm via indwelling heparin-anticoagulated IV catheters, or by venipunctures at 0 (baseline), 2, 5, 7.5, 10, 12.5, 15, 20, 25, 30, 45, 60, 90, 120, 240, and 360 minutes post-dose in each treatment period and were analyzed using an established analysis method. Tmax is the amount of time it takes for epinephrine to reach peak concentration in plasma during the treatment period.
Time Frame: Pre-dose to 6 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: min
Arm/Group | Treatment T | Treatment C
Number analyzed (Participants) | 23 | 23
min | 2.3 (1.7) | 3.4 (4.3)

5. Primary Outcome: Half-life (t1/2) of Total Epinephrine
Description: Patient PK blood samples were taken from a vein in a hand or arm via indwelling heparin-anticoagulated IV catheters, or by venipunctures at 0 (baseline), 2, 5, 7.5, 10, 12.5, 15, 20, 25, 30, 45, 60, 90, 120, 240, and 360 minutes post-dose in each treatment period and were analyzed using an established analysis method. Half-life (t1/2) is the amount of time it takes for epinephrine to decrease to half the peak concentration in plasma during the treatment period.
Time Frame: Pre-dose to 6 hours post-dose
Population: as for outcome 2
Measure: Mean (Full Range); unit: min
Arm/Group | Treatment T | Treatment C
Number analyzed (Participants) | 23 | 23
min | 145.9 [1.7 to 864.0] | 289.8 [1.8 to 1996.3]

6. Primary Outcome: Concentration vs. Time for Total Epinephrine From Time Zero to 6 Hours Post-dose
Description: Patient PK blood samples were taken from a vein in a hand or arm via indwelling heparin-anticoagulated IV catheters, or by venipunctures at 0 (baseline), 2, 5, 7.5, 10, 12.5, 15, 20, 25, 30, 45, 60, 90, 120, 240, and 360 minutes post-dose in each treatment period and were analyzed using an established analysis method.
Time Frame: Pre-dose to 6 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Treatment T | Treatment C
Number analyzed (Participants) | 23 | 23
pg/mL
  0 min (Baseline) | 2.6 (8.7) | 4.3 (16.7)
  2 min post-dose | 861.5 (528.2) | 189.0 (123.3)
  5 min post-dose | 379.4 (203.0) | 99.1 (67.0)
  7.5 min post-dose | 186.6 (97.7) | 48.8 (30.0)
  10 min post-dose | 118.3 (65.8) | 39.7 (22.9)
  12.5 min post-dose | 75.6 (42.2) | 33.9 (21.4)
  15 min post-dose | 46.8 (41.7) | 32.0 (23.3)
  20 min post-dose | 22.9 (21.3) | 30.1 (19.8)
  25 min post-dose | 10.9 (19.9) | 20.3 (17.9)
  30 min post-dose | 10.5 (16.1) | 17.7 (19.4)
  45 min post-dose | 10.5 (22.5) | 19.8 (21.2)
  60 min post-dose | 8.7 (13.9) | 13.2 (14.5)
  90 min post-dose | 3.5 (9.4) | 11.2 (18.2)
  120 min post-dose | 6.5 (13.2) | 6.9 (12.0)
  240 min post-dose | 16.1 (23.8) | 17.7 (17.6)
  360 min post-dose | 17.1 (23.9) | 17.2 (20.4)

ADVERSE EVENTS:
Time Frame: Throughout entire study period
Arm/Group | Treatment T | Treatment C
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 1/23 | 2/23
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment T (N=23) | Treatment C (N=23)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Viral Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other